CLINICAL TRIAL: NCT06633198
Title: Heat, Microvascular Function and Aging
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Hughes (Other)
Responsible Party: Sponsor-Investigator, William Hughes, Assistant Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO00052867
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-04

CONDITIONS: Aging
Keywords: Passive heating; Aging; Microvascular; Autophagy
MeSH Terms: interventions — NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Passive Heating of lower limbs (Experimental): The lower limbs will be immersed in warm circulating water for 60 minutes.
  Interventions: Procedure: Passive Heating; Drug: L-NAME

INTERVENTIONS:
Procedure: Passive Heating — The lower limbs will be immersed in warm (42C) circulating water for 60 minutes.
Drug: L-NAME — L-NAME will be used during measurement of cutaneous microvascular function to test the dependency upon NO to elicit vasodilation.

SUMMARY:
Vascular dysfunction is a common factor in many chronic debilitating diseases, contributing to morbidity and mortality. With the onset of chronic disease or exposure to stress, the vasculature displays an inability to adequately respond to increased blood flow demands, manifesting in a reduced ability or altered mechanism of vasodilation. Aging is an independent risk factor in the development of cardiovascular disease, and reduces vasodilator capacity, or alters the mechanism by which vasodilation occurs in multiple vascular beds. Chronic exercise/physical activity is one of the most potent ways to enhance vascular function, resulting in favorable outcomes such as reductions in blood pressure, and improved ability to perform activities of daily living. Barriers to exercise or failure of long-term adherence preclude many populations from the cardiovascular benefits of exercise, thus further enhancing cardiovascular risk. Avenues to mimic blood flow patterns observed with exercise may exert beneficial effects without the need for the ability to exercise. Recent evidence has demonstrated that passive heat therapy, or chronic heat exposure (~ +1°C in core temperature) results in reductions in major adverse cardiovascular events, blood pressure and improved large artery endothelial function, primarily through preservation of large artery function in response to vascular stress. It is unclear whether microvascular function is augmented in response to acute heat exposure, or whether this can protect against vascular insults particularly in older adults. Some preliminary evidence in humans suggest that autophagy, a cell recycling process is involved in the beneficial cardiovascular effects, as short-term heat exposure upregulates markers of autophagy. Previous evidence from our lab indicates that autophagy governs the mechanism by which microvascular vasodilation occurs. The role of autophagy in mediating the beneficial effects of passive heating is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18-80 yrs. of age
* No more than 1 cardiovascular risk factor (see list in exclusion criteria)

Exclusion Criteria:

* Cardiovascular Risk Factors
* Uncontrolled/unmanaged hypertension and/or use of current anti-hypertensive therapy
* Current Tobacco product use or within last 6 months
* BMI greater than 30
* Hyperlipidemia - diagnosed and/or taking medications to manage
* Hypercholesterolemia - diagnosed and/or taking medications to manage (e.g. statins)
* Type 1 or Type 2 Diabetes
* Use of anti-coagulant or anti-platelet drugs
* Use of beta blockers
* Symptomatic coronary artery disease
* Diagnosed Heart Failure (Any classification above Class I as defined by NY Heart Association)
* Diagnosed renal impairment Renal impairment defined, according to National Kidney Foundation as abnormalities of kidney structure or function, present for greater than 3 months, including:
* Albuminuria (ACR ≥ 30 mg/g)
* Urine sediment abnormalities
* Electrolyte and other abnormalities due to tubular disorders
* Structural abnormalities detected by imaging
* History of kidney transplantation
* Decreased glomerular filtration rate (GFP < 60 mL/min/1.73 m2)
* Current Hormone Replacement Therapy Use
* History of retinopathy
* Documented neuromuscular disorders
* Porphyria Cutanea Tarda (blistering of skin to sun; photosensitivity)
* Pregnancy (Young Female subjects)
* Allergies to povidone iodine
* Tattoos on lower arm (forearm)
* Use of erectile dysfunction medication in the past 6 months
* Use of topical/non-topical steroids in last 6 months (e.g. cortisone cream)
* Active anti-cancer treatment or treatment within last 12 months
* Active COVID-19 or within the past 3 months
* Gender Reassignment Therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cutaneous microvascular function | Baseline, 60 minutes post I/R, and 60 minutes post hot water immersion + I/R injury
  Change in cutaneous microvascular function assessed via microdialysis infusion of acetylcholine (dose response) in the presence and absence of L-NAME to test the dependency upon NO to elicit vasodilation.

SECONDARY OUTCOMES:
Spontaneous baroreflex sensitivity | Baseline, 60 minutes post I/R, 60 minutes post hot water immersion + I/R injury
  Change in spontaneous BRS
24-hour (Ambulatory) Blood Pressure | Baseline
  Ambulatory blood pressure (systolic, diastolic) for both peripheral and aortic blood pressure
Change in plasma concentration of heat shock proteins | Baseline and 60 minutes post hot water immersion
  Change in the plasma concentrations of various heat shock proteins (HSP 70, 90)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided